CLINICAL TRIAL: NCT00132171
Title: High Eradication Rates of Helicobacter Pylori With a New Sequential Treatment
Brief Title: Helicobacter Pylori Eradication With a New Sequential Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 66/2000/J
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Helicobacter Pylori Infection; Non Ulcer Dyspepsia; Duodenal Ulcer; Gastric Ulcer; Chronic Active Gastritis; Gastritis
Keywords: Helicobacter pylori; Eradication; Sequential therapy; Standard therapy
MeSH Terms: conditions — Duodenal Ulcer; Stomach Ulcer; Gastritis

INTERVENTIONS:
Drug: Sequential therapy

SUMMARY:
Eradication rates of Helicobacter pylori (H. pylori) with standard triple therapy are disappointing, and studies from several countries confirm this poor performance. The study aimed to assess the eradication rate of a new sequential treatment regimen compared with conventional triple therapy for the eradication of H. pylori infection.

DETAILED DESCRIPTION:
One thousand and forty-nine dyspeptic patients were studied prospectively. H. pylori-infected patients were randomized to receive 10-day sequential therapy [rabeprazole (20 mg twice daily) plus amoxicillin (1 g twice daily) for the first 5 days, followed by rabeprazole (20 mg), clarithromycin (500 mg) and tinidazole (500 mg, all twice daily for the remaining 5 days] or standard 7-day therapy [corrected] [rabeprazole (20 mg), clarithromycin (500 mg) and amoxicillin (1 g), all twice daily]. H. pylori status was assessed by histology, rapid urease test and 13C-urea breath test at baseline and 6 weeks or more after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of active H. pylori infection
* Age >18 years

Exclusion Criteria:

* Allergy to drug administered
* Liver or kidney failure
* Pregnancy
* Previous treatment for H. pylori infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2001-01; Study Completion 2001-12

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate

SECONDARY OUTCOMES:
Compliance to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Zullo, MD, Principal Investigator — Nuovo Regina Margherita Hospital
Locations (1):
- Gastroenterology - Nuovo Regina Margherita Hospital, Rome, Italy

REFERENCES:
- [Result] Zullo A, Vaira D, Vakil N, Hassan C, Gatta L, Ricci C, De Francesco V, Menegatti M, Tampieri A, Perna F, Rinaldi V, Perri F, Papadia C, Fornari F, Pilati S, Mete LS, Merla A, Poti R, Marinone G, Savioli A, Campo SM, Faleo D, Ierardi E, Miglioli M, Morini S. High eradication rates of Helicobacter pylori with a new sequential treatment. Aliment Pharmacol Ther. 2003 Mar 1;17(5):719-26. doi: 10.1046/j.1365-2036.2003.01461.x. PMID 12641522